CLINICAL TRIAL: NCT06111729
Title: Habit Awareness Device for Treatment of Onychophagia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-12025533
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Nail Biting
MeSH Terms: conditions — Nail Biting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- HabitAware Participants (Experimental): Patients will be asked to wear the HabitAwareness bracelet for 12 weeks. The bracelet provides the attention stimulus of gentle vibration when the motion of nail biting is sensed.
  Interventions: Device: HabitAware group

INTERVENTIONS:
Device: HabitAware group — A device that provides gentle vibration when the motion of nail biting is sensed will be provided to all participants. Participants will use an app that connects to the device to track the frequency of their nail biting over the study period.

SUMMARY:
This clinical trial wants to find out if using a special bracelet that vibrates gently whenever someone with a nail-biting problem bites their nails can help them stop. The investigators are looking at adults who bite their nails a lot. If this bracelet works, it could make nail-biters bite their nails less and have a better life.

The main question the investigators are trying to answer is: "Does the gentle vibration from the bracelet make people bite their nails less?"

The investigators will give participants a bracelet that vibrates when it senses nail-biting for 12 weeks. Participants will need to download an app that connects to the bracelet. This app will help the investigators keep track of how often participants get these vibration signals and see if nail-biting decreases while using the bracelet.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with onychophagia
2. Must understand and voluntarily sign an informed consent form
3. Must be aged 18-95 years at the time of consent
4. Must be able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Subject is unable to provide written informed consent for any reason.
2. Subject is sensitive or allergic to any of the elements included in this study.
3. Subject is unable to complete the required pain dairy.
4. Subject is pregnant, planning pregnancy, or nursing.
5. Subject does not have a compatible personal device with either IOS 13.0 or greater or Android version 6.0 or greater.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Nail Biting Behavior as Measured by Number of Patient Reported Vibrations a Day | baseline; 4 weeks; 8 weeks; 12 weeks

SECONDARY OUTCOMES:
Change in nail length in millimeters | Monthly for 3 months
Change in nail health as measured by Malone-Massler Scale For Nail Biting | baseline; 3 months
  The lowest score is 0 meaning nails not bitten, free margin intact; the highest score is 3+ meaniing nails are severely bitten, fingernails bitten beyond free edge; nail margin below soft tissue border

CONTACTS AND LOCATIONS:
Overall Officials: Shari Lipner, MD, PhD, Principal Investigator — Professor of Clinical Dermatology
Locations (1):
- Weill Cornell Department of Dermatology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification
Supporting Information: SAP, CSR
Time Frame: Immediately following publication. no end date
Access Criteria: Anyone who wishes to access the data

REFERENCES:
- [Background] Stiede JT, Woods DW, Idnani AK, Pritchard J, Klobe K, Kumar S. Pilot trial of a technology assisted treatment for trichotillomania. J Obsessive Compuls Relat Disord. 2022 Apr;33:100726. doi: 10.1016/j.jocrd.2022.100726. Epub 2022 Apr 29. PMID 37305101